CLINICAL TRIAL: NCT00318682
Title: Evaluation and Medico Economic Study of FIBROSCAN in Patients With Viral Hepatitis
Brief Title: Evaluation and Medico-Economic Study of FIBROSCAN in Patients With Viral Hepatitis
Acronym: FIBROSTIC
Status: Terminated | Type: Observational
Why Stopped: enough patients have been enrolled for the statistic analysis
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Mathieu QUINTIN, Department Clinical Research of Developpement
Other Study IDs: IC0504
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis, Viral, Human
Keywords: biopsy; FIBROSCAN
MeSH Terms: conditions — Hepatitis, Viral, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biological samples to evaluate the hepato-fibrosis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FIBROSCAN — diagnostic examination of the hepato fibrosis

SUMMARY:
A new approach to the evaluation of liver fibrosis has been proposed using PULSOMETRY. The objective is to evaluate the diagnostic performances of the FIBROSCAN technique, together with non-invasive techniques, and to determine how it is able to predict the histological fibrosis score, defined by the METAVIR score. This transversal study aims to compare the evaluation of hepatic fibrosis obtained by FIBROSCAN and histology (METAVIR score) in 2550 consecutive patients taken in charge for a liver biopsy. The results of the study will compare the respective performances of these techniques in the prediction of the METAVIR score, and help in the recommendation of the care of patients with viral hepatitis B and C; these methods will undergo a medico-economic study.

DETAILED DESCRIPTION:
The gold standard for the evaluation of fibrosis is considered as the METAVIR score by the clinicians. The results of this score are currently used for clinical decisions and description of the evolution of the disease. FIBROSCAN would be interesting in avoiding liver biopsies, if it was able to predict accurately the METAVIR score obtained if a liver biopsy was performed. The data available on diagnostic performances of FIBROSCAN are incomplete, the number of patients studied and the methods selection (blindness of the results of other techniques) are not precise in some of them. The main objective of this study is therefore to evaluate the performance of FIBROSCAN in the prediction of METAVIR score > 2 (vs F0 or F1). An ancillary study will try to evaluate the diagnostic performance of FIBROSCAN in the global prediction of METAVIR score. A statistical method will be tested using the reference method as an ordinal polytropic variable. Half of the sample (1250 patients) will be used to determine the best THERSHOLD of FIBROSCAN in each of the clinical subgroups of patients, in order to obtain a high sensibility. The second half will be used as the validation sample, and the threshold will be used to estimate the sensibility, specificity and other diagnostic parameters of the FIBROSCAN. The secondary objectives are:

1. to evaluate the performance of FIBROSCAN in the prediction of METAVIR score in adjacent classes of fibrosis (F0-F1, F1-F2, F2-F3, F3-F4), and
2. to study the association between elastometry and fibrosis surface obtained by morphometry (considered as the best evaluation of global liver fibrosis).

This technique will be applied to a restricted number of biopsies (consecutive biopsies > 2cm).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B or C
* With liver biopsy indication
* Patient information

Exclusion Criteria:

* Drug hepatitis
* Metabolic hepatology
* Steatosis or non-alcoholic steatohepatitis
* Autoimmune hepatopathy
* Non-contraindication to liver biopsy
* Non-contraindication to FIBROSCAN examination
* Ascites
* Obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with hepatitis B or C
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Degos, PhD, Principal Investigator — Hopital Beaujon
Locations (2):
- France (2):
  - Hopital Beaujon, Clichy
  - Hopital Saint-Antoine, Paris